CLINICAL TRIAL: NCT06855004
Title: Prospective Multicenter Cohort of Patients With Fibrosing Interstitial Lung Disease Admitted to Intensive Care or Critical Care Units for Acute Respiratory Failure
Brief Title: Prospective Cohort of Patients With Fibrosing Interstitial Lung Disease Admitted for Acute Respiratory Failure
Acronym: PIDREA
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP241343
Record Dates: First submitted 2025-02-12; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-12

CONDITIONS: Fibrosing Interstitial Lung Disease
Keywords: fibrosing interstitial lung disease; intensive care or critical care units; mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective, multicenter study focuses on patients with fibrosing interstitial lung diseases (ILD) admitted to intensive care units (ICUs) for acute respiratory failure (ARF). ILD encompasses a group of heterogeneous disorders characterized by progressive fibrotic and inflammatory damage to the lung interstitium, often resulting in chronic respiratory failure. Acute respiratory failure in these patients is a severe and frequent complication caused by various factors, including infections, pulmonary embolism, cardiac decompensation, or acute exacerbation of fibrosis. Despite advances in treatment, ICU management of these patients remains a clinical and ethical challenge due to high mortality rates and limited evidence-based guidance.

The study's primary objective is to assess 6-month survival following ICU admission for ARF in ILD patients. Secondary objectives include identifying prognostic factors for mortality, characterizing ICU and hospital mortality rates, and evaluating the use of organ support measures (e.g., oxygen therapy, invasive or non-invasive mechanical ventilation). Additionally, the study will examine the frequency of lung transplantation, acquired ICU infections, and decisions to limit or withdraw life-sustaining therapies.

Importantly, this research aims to address a significant gap in current knowledge by building a large, descriptive, prospective cohort of ILD patients. A critical aspect of the study is the evaluation of patients' quality of life (QoL) six months after ICU discharge, using a dedicated questionnaire. This information will provide essential insights into the long-term benefits of ICU care for these patients, complementing survival data with QoL outcomes to better guide clinical decision-making and improve patient-centered care.

DETAILED DESCRIPTION:
Fibrosing interstitial lung disease (ILD) encompasses a number of heterogeneous pathologies that share the common features of fibrotic and inflammatory lesions of the lung parenchyma, particularly in the space between the lung epithelium and endothelium. An epidemiological study carried out in France in the Seine Saint Denis département (PID93) estimates the prevalence of all PIDs combined at 97/100,000. Despite recent advances, ILD classically evolves towards chronic end-stage respiratory failure. Acute respiratory failure in the context of ILD is a common and severe complication, often necessitating intensive care for specialized ventilatory support.

The causes of acute respiratory failure in patients with ILD are varied. They include community-acquired or opportunistic infections (in patients on immunosuppressive therapy), pulmonary embolism and cardiac decompensation. Acute exacerbation of pulmonary fibrosis is a sudden worsening of respiratory function characterized by rapid-onset hypoxemia and new bilateral pulmonary infiltrates on imaging, often occurring without a clear cause. It involves acute lung injury superimposed on underlying fibrotic lung disease, typically associated with a high mortality rates at 3 months estimated at 50%, and 90% in patients requiring invasive mechanical ventilation. This complication occurs most frequently in advanced idiopathic pulmonary fibrosis (IPF), with an annual incidence of between 5% and 10%.

Current management guidelines for fibrosing interstitial lung diseases (ILDs) are primarily based on outdated, retrospective, single-center studies. The latest recommendations for idiopathic pulmonary fibrosis (IPF) (ATS 2022) suggest transferring patients to intensive care in cases of acute exacerbations when lung transplantation is planned, a reversible cause of deterioration is identified, or etiological investigations remain incomplete. However, in practice, acute respiratory failure in this context presents both clinical and ethical challenges due to the limited benefits of invasive mechanical ventilation for most patients with fibrosing ILDs.

Recent advancements have influenced patient care: the incidence of fibrosing ILDs has increased, partly due to improved diagnostic approaches; anti-fibrotic therapies have become the standard of care, slowing disease progression; and advances in protective ventilation and high-flow oxygen therapy have encouraged more active involvement from intensivists. Additionally, the development of extracorporeal membrane oxygenation (ECMO) in awake patients and super-emergency lung transplantation has expanded intensive care options for these patients.

The prognosis for patients with ILD admitted to intensive care remains poor. French studies by Gaudry et al. and Tandjaoui et al. highlight the unfavorable outcomes in approximately 100 patients, primarily with IPF and non-specific interstitial pneumonias, particularly when invasive mechanical ventilation is required. International literature provides limited guidance due to heterogeneous and often undocumented fibrosis etiologies in available retrospective single-center studies.

In summary, personalized, multidisciplinary care by expert teams is crucial for improving outcomes. The concentration of cases at specialized centers hinders the establishment of large prospective cohorts, leaving intensive care teams without robust, up-to-date data on diagnostics and treatments. To address these gaps, we aim to create a large, descriptive, prospective cohort across multiple centers and evaluate patients' quality of life six months post-intensive care using a dedicated questionnaire. These insights are essential for assessing the comprehensive benefits of intensive care stays.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalization in intensive care for acute respiratory failure
2. Requirement for standard oxygen therapy with an O2 flow rate > 6 l/min, high-flow oxygen therapy, or mechanical ventilation (non-invasive or invasive)
3. Age ≥ 18 years
4. Patient (male or female) with chronic interstitial lung disease (ILD)

   1. Diagnosis of chronic ILD confirmed by a multidisciplinary discussion (MDD) prior to admission to intensive care, or
   2. Diagnosis of chronic ILD made during the intensive care stay due to the acute episode and confirmed by an expert opinion.

Exclusion Criteria:

1. Patient under legal guardianship or with restricted freedom
2. Patient hospitalized for psychiatric reasons or with a severe psychiatric illness causing a disability, subject to legal protection measures
3. Pregnant woman
4. Patient already enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a heterogeneous patient population requiring specialized expertise, and their prognosis in intensive care is poor without effective curative treatment. To date, there are no prospective multicenter studies in intensive care targeting this population. Additionally, there is no data on their quality of life following an intensive care stay.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2030-07-28 (Estimated); Study Completion 2030-10-28 (Estimated)

PRIMARY OUTCOMES:
Overall survival at 6 months. | 6 months
  Survival will be assessed from the date of admission to intensive care (Day 0) until the date of death from any cause. Patients who are lost to follow-up or alive at the end of their follow-up period will be censored on the last date their status was documented. The maximum follow-up duration for each patient will be six months. For patients lost to follow-up before the planned follow-up period ends, their vital status (alive or deceased) will be verified with their town of birth registry.

SECONDARY OUTCOMES:
Overall survival in the intensive care unit (ICU) and hospital | Up to 6 months
Length of stay in the ICU and hospital | Up to 6 months
Percentage of patients requiring non-invasive ventilation techniques (e.g., high-flow oxygen therapy, non-invasive ventilation) | Up to 6 months
Percentage of patients requiring invasive ventilation techniques or extracorporeal membrane oxygenation (ECMO) | Up to 6 months
Percentage of patients requiring catecholamine infusion | Up to 6 months
Percentage of patients requiring renal replacement therapy | Up to 6 months
Percentage of patients urgently listed for lung transplantation and/or undergoing lung transplantation during hospitalization | Up to 6 months
Percentage of patients with at least one ICU-acquired infection | Up to 6 months
  Percentage of patients with at least one ICU-acquired infection, including:
  * Ventilator-associated pneumonia (defined by clinical symptoms and microbiological evidence: >10⁶ colony forming unit (CFU)/mL in tracheal aspirates, >10⁴ colony forming unit (CFU)/mL in bronchoalveolar lavage fluid, or >10³ colony forming unit (CFU)/mL in protected distal samples)
  * Bacteremia (catheter-related or of unknown origin)
  * Fungemia (catheter-related or of unknown origin)
  * Viral infections requiring systemic antiviral treatment
Percentage and timing of decisions to limit active therapeutic interventions | Up to 6 months
Barthel Index at 6 months | Admission date (D0) and 6 months
  Barthel Index at 6 months (assessed via phone)
Percentage of patients dependent on long-term oxygen therapy at 6 months | 6 months
Quality of life score (SF-36) before and after intensive care | Admission date (D0) and 6 months
  Quality of life score (SF-36) before ICU admission and at 6 months post-ICU

CONTACTS AND LOCATIONS:
Overall Officials: Nathan EBSTEIN, Dr, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Avicenne APHP Réanimation médico-chirurgicale, Bobigny, France

IPD SHARING:
Plan to Share IPD: No